CLINICAL TRIAL: NCT01884350
Title: Assessment of an Education and Guidance Programme for Eliquis Adherence in Non-Valvular Atrial Fibrillation (AEGEAN)
Acronym: AEGEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CV185-220; 2013-000055-41 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-24 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Non-valvular Atrial Fibrillation
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Apixaban (Primary SOC information) (Experimental): Apixaban 2.5 mg or 5 mg by mouth twice daily for 48 weeks and Primary Standard of Care (SOC) information
  Interventions: Drug: Apixaban
- Arm 2: Apixaban (Additional Educational Program) (Experimental): Apixaban 2.5 mg or 5 mg by mouth twice daily for 48 weeks and Additional Educational Program
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis; BMS-562247

SUMMARY:
The study purpose is to assess the impact of an educational program on patient adherence in patients taking Apixaban for SPAF at 24 weeks

DETAILED DESCRIPTION:
SPAF=Stroke Prevention in Atrial Fibrillation

ISTH=International Society on Thrombosis and Hemostasis

Primary Purpose: Other: To measure adherence to the study medication using an electronic monitoring device over the first 24 weeks on study medication

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosed non-valvular Atrial Fibrillation (AF) or atrial flutter (documented by 12-lead electrocardiogram (ECG) or Holter recording) and eligible for oral anticoagulant (OAC) therapy
2. Presence of at least one of the following risk factors for stroke:

   Prior stroke or transient ischaemic attack (TIA)
   * Age ≥75 years
   * Hypertension
   * Diabetes mellitus
   * Symptomatic heart failure [New York Heart Association (NYHA) Class ≥II]
3. Must be able to self-administer treatment
4. Either Vitamin K antagonists (VKA) treated or VKA naive. Patients treated with VKA should have received the VKA treatment for ≥3 months. VKA naïve patients should not have received VKA treatment for more than 30 days within the last 12 months. Patients who are not described by either of the above criteria are not eligible for the study
5. Patients previously treated with acetylsalicylic acid (ASA) for stroke prevention are allowed (and will switch to Apixaban)
6. Patients with screening mini-mental state examination (MMSE) more than 24
7. Subject Re-enrollment: This study does not permit the re-enrollment of a subject that has discontinued the study as a pre-treatment failure

Age and Reproductive Status:

* i) Men and women ≥18 years of age
* ii) Women of childbearing potential (WOCBP) must use method(s) of contraception based on the tables in protocol. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study medication
* iv) Women must not be breastfeeding
* v) Men who are sexually active with women of childbearing potential (WOCBP) must use any contraceptive method with a failure rate of less than 1% per year
* vi) Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile); and azoospermic men do not require contraception

Exclusion Criteria:

1. Target Disease Exceptions:

   1. Atrial fibrillation or flutter due to reversible causes (e.g. thyrotoxicosis, pericarditis)
   2. Clinically significant (moderate or severe) mitral stenosis
   3. Cardiac valvular disease requiring surgery
   4. Planned major surgery or/and invasive procedure and/or atrial fibrillation or flutter, ablation procedure and/or cardioversion
   5. Patients receiving Rivaroxaban, Dabigatran or Apixaban
2. Medical History and Concurrent Diseases:

   1. Conditions other than atrial fibrillation that require chronic anticoagulation (e.g., prosthetic mechanical heart valve, venous thromboembolism; also see Section 3.4, Concomitant Treatments)
   2. Patient with serious bleeding in the last 6 months or with a lesion or condition at high risk of bleeding such as:

      * Active peptic ulcer disease, current or recent gastrointestinal ulceration
      * Known or suspected esophageal varices
      * Recent ischemic stroke (within 7 days)
      * Recent brain or spinal injury or intracranial hemorrhage
      * Recent brain, spinal or ophthalmic surgery
      * Arteriovenous malformations
      * Vascular aneurysms
      * Major intraspinal or intracerebral vascular abnormalities
      * Documented hemorrhagic tendencies or blood dyscrasias
      * Presence of malignant neoplasms at high risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2013-10-15 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (186):
- Belgium (13):
  - Local Institution, Antwerp
  - Local Institution, Arlon
  - Local Institution, Bonheiden
  - Local Institution, Braine-l'Alleud
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Gilly
  - Local Institution, Hasselt
  - Local Institution, Leuven
  - Local Institution, Liège
  - Local Institution, Ronse
  - Local Institution, Woluwe-Saint-Lambert
  - Local Institution, Yvoir
- France (55):
  - Local Institution, Saint-Etienne, Cedex 2
  - Local Institution, Abbeville
  - Local Institution, Aix-en-Provence
  - Local Institution, Avignon
  - Local Institution, Bayonne
  - Local Institution, Béziers
  - Local Institution, Bobigny
  - Local Institution, Bordeaux
  - Local Institution, Boulogne-Billancourt
  - Local Institution, Brest
  - Local Institution, Bron
  - Local Institution, Caen
  - Local Institution, Cambrai
  - Local Institution, Cannes
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Chartes
  - Local Institution, Châtellerault
  - Local Institution, Cholet
  - Local Institution, Clermont-Ferrand
  - Local Institution, Colombes
  - Local Institution, Corbeil-Essonnes
  - Local Institution, Créteil
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Haguenau
  - Local Institution, La Rochelle
  - Local Institution, Le Chesnay
  - Local Institution, Lille
  - Local Institution, Longjumeau
  - Local Institution, Marseille
  - Local Institution, Montfermeil
  - Local Institution, Montpellier
  - Local Institution, Nantes
  - Local Institution, Neuilly-sur-Seine
  - Local Institution, Nice
  - Local Institution, Nîmes
  - Local Institution, Orléans
  - Local Institution, Paris
  - Local Institution, Pau Universite Cedex
  - Local Institution, Pessac
  - Local Institution, Plan-de-Cuques
  - Local Institution, Rennes
  - Local Institution, Saint-Benoît
  - Local Institution, Saint-Denis
  - Local Institution, Salouël
  - Local Institution, Sète
  - Local Institution, Strasbourg
  - Local Institution, Thionville
  - Local Institution, Thonon-les-Bains
  - Local Institution, Toulouse
  - Local Institution, Tourcoing
  - Local Institution, Valence
  - Local Institution, Valenciennes
  - Local Institution, Vesoul
  - Local Institution, Wardenburg
- Germany (55):
  - Local Institution, Spaichingen, Baden-wurttembe
  - Local Institution, Krombach, Bavaria
  - Local Institution, Augsburg
  - Local Institution, Aurich
  - Local Institution, Bad Homburg
  - Local Institution, Balingen
  - Local Institution, Bamberg
  - Local Institution, Berin
  - Local Institution, Berlin
  - Local Institution, Chemnitz
  - Local Institution, Deggingen
  - Local Institution, Dillingen
  - Local Institution, Dresden
  - Local Institution, Erfurt
  - Local Institution, Essen
  - Local Institution, Flörsheim
  - Local Institution, Friedberg
  - Local Institution, Gars/Inn
  - Local Institution, Göttingen
  - Local Institution, Grossheirath Rossbach
  - Local Institution, Hamburg
  - Local Institution, Haßloch
  - Local Institution, Heidelberg
  - Local Institution, Heidenau
  - Local Institution, Kassel
  - Local Institution, Kelkheim
  - Local Institution, Künzing
  - Local Institution, Langestrasse
  - Local Institution, Leipzig
  - Local Institution, Lollar
  - Local Institution, Ludwigsburg
  - Local Institution, Mammendorf
  - Local Institution, Mannheim
  - Local Institution, Markkleeberg
  - Local Institution, Münster
  - Local Institution, Myen
  - Local Institution, Neukirchen
  - Local Institution, Neunirchen
  - Local Institution, Northeim
  - Local Institution, Obermichelbach
  - Local Institution, Papenburg
  - Local Institution, Pirna
  - Local Institution, Riesa
  - Local Institution, Rodgau
  - Local Institution, Rotenburg /fulda
  - Local Institution, Sinzheim
  - Local Institution, Stockach
  - Local Institution, Unterschneidheim
  - Local Institution, Wallerfing
  - Local Institution, Wangen
  - Local Institution, Weißenhorn
  - Local Institution, Wermsdorf
  - Local Institution, Wetzlar
  - Local Institution, Weyhe
  - Local Institution, Winsen
- Italy (27):
  - Local Institution, Milan, MI
  - Local Institution, Arezzo
  - Local Institution, Bologna
  - Local Institution, Castelfranco Veneto (tv)
  - Local Institution, Catanzaro
  - Local Institution, Cremona
  - Local Institution, Florence
  - Local Institution, Foggia
  - Local Institution, L’Aquila
  - Local Institution, Mestre
  - Local Institution, Milan
  - Local Institution, Naples
  - Local Institution, Napoli
  - Local Institution, Palermo
  - Local Institution, Pavia
  - Local Institution, Perugia
  - Local Institution, Piacenza
  - Local Institution, Reggio Emilia
  - Local Institution, Roma
  - Local Institution, San Daniele Del Friuli(udine)
  - Local Institution, Siena
  - Local Institution, Torino
  - Local Institution, Treviso
  - Local Institution, Varese
  - Local Institution, Vicenza
  - Local Institution, Vimercate
  - Local Institution, Viterbo
- Spain (13):
  - Local Institution, San Sebastián de los Reyes, Madrid
  - Local Institution, Aldaia
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Galdakao
  - Local Institution, Madrid
  - Local Institution, Murcia
  - Local Institution, Oviedo
  - Local Institution, Santiago de Compostela
  - Local Institution, Tarragona
  - Local Institution, Valencia
  - Local Institution, Viladecans
  - Local Institution, Zaragoza
- Switzerland (6):
  - Local Institution, Lugano, Canton Ticino
  - Local Institution, Fribourg, Canton
  - Local Institution, Baden
  - Local Institution, Bern
  - Local Institution, Winterthur
  - Local Institution, Zurich
- United Kingdom (17):
  - Local Institution, Craigavon, Armagh
  - Local Institution, Darlington, County Durham
  - Local Institution, Exeter, Devon
  - Local Institution, Bournemouth, Dorset
  - Local Institution, Poole, Dorset
  - Local Institution, Westcliff-on-Sea, Essex
  - Local Institution, Ashford, KENT
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Airdrie, Lancashire
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Stoke-on-Trent, Staffordshire
  - Local Institution, Birmingham, WEST Midlands
  - Local Institution, Dudley, WEST Midlands
  - Local Institution, Hereford
  - Local Institution, Oldham
  - Local Institution, Somerset
  - Local Institution, Tauton

REFERENCES:
- [Derived] Montalescot G, Brotons C, Cosyns B, Crijns HJ, D'Angelo A, Drouet L, Eberli F, Lane DA, Besse B, Chan A, Vicaut E, Darius H; AEGEAN Study Investigators. Educational Impact on Apixaban Adherence in Atrial Fibrillation (the AEGEAN STUDY): A Randomized Clinical Trial. Am J Cardiovasc Drugs. 2020 Feb;20(1):61-71. doi: 10.1007/s40256-019-00356-2. PMID 31243691
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1217 participants were enrolled, 1162 randomized (583 Primary SOC,579 AEP). 55 were enrolled but not randomized. Of the 55, 13 no longer met study criteria, 13 withdrew consent, 3 lost to follow-up, 10 other and 16 unknown.
Groups:
- Apixaban (Primary SOC): Participants were treated with Apixaban 2.5 mg or 5 mg by mouth twice daily for 48 weeks and received Primary Standard of Care (SOC) information.
- Apixaban (Additional Educational Program): Participants were treated with Apixaban 2.5 mg or 5 mg by mouth twice daily for 48 weeks and received the Additional Educational Program (AEP). After the initial 24-week primary endpoint period, participants in the AEP group were randomized 1:1 to continue receiving AEP or stop receiving AEP and revert to Standard of Care (SOC) information via the Apixaban (Secondary SOC) group.
- Apixaban (Secondary SOC): Participants were originally in the Apixaban (AEP) arm and treated with Apixaban 2.5 mg or 5 mg by mouth twice daily and Additional Educational Program (AEP) for the first 24 weeks. After the initial 24-week primary endpoint period participants stopped receiving AEP and were transferred from Apixaban (AEP) arm, stopped the Additional Educational Program (AEP), and switched to the Standard of Care (SOC) information for an additional 24 weeks.
Period: Primary Efficacy Analysis Set (24 Weeks)
Arm/Group | Apixaban (Primary SOC) | Apixaban (Additional Educational Program) | Apixaban (Secondary SOC)
Started (Primary Efficacy Analysis set: All randomized patients.) | 583 | 579 | 0 (Participants were not randomized to this arm until after initial 24-week period)
Safety Analysis Set (All randomized patients who received any study drug.) | 604 | 558 | 0
Completed | 529 | 525 | 0
Not Completed | 54 | 54 | 0
Not completed — Subject Withdrew Consent | 17 | 20 | 0
Not completed — Death | 6 | 4 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Serious Adverse Event | 7 | 6 | 0
Not completed — Adverse Event | 15 | 11 | 0
Not completed — Drug Interruption >30 Consecutive Days | 0 | 2 | 0
Not completed — Inclusion/exclusion criterion | 2 | 5 | 0
Not completed — Helping Hand not used | 2 | 0 | 0
Not completed — Helping Hand not used, treatment taken | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Medical reason | 3 | 3 | 0
Period: Primary Efficacy Analysis Set (48 Weeks)
Arm/Group | Apixaban (Primary SOC) | Apixaban (Additional Educational Program) | Apixaban (Secondary SOC)
Started (Primary Efficacy Analysis Set. 1 completed initial period but was not rand. to 2nd 24-week period) | 583 | 263 (After 24 weeks participants were randomized to continue AEP or stop AEP and revert to SOC.) | 261 (After 24 weeks participants were randomized to continue AEP or stop AEP and revert to SOC.)
Safety Analysis Set (All randomized patients who received any study drug.) | 604 | 308 | 223
Completed | 503 | 250 | 250
Not Completed | 80 | 13 | 11
Not completed — Subject Withdrew Consent | 21 | 0 | 2
Not completed — Death | 7 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Serious Adverse Event | 17 | 6 | 3
Not completed — Adverse Event | 17 | 3 | 0
Not completed — Drug Interruption >30 Consecutive Days | 3 | 0 | 2
Not completed — Helping Hand not used | 4 | 0 | 0
Not completed — Helping Hand not used, treatment taken | 3 | 0 | 0
Not completed — Medical reason | 4 | 1 | 0
Not completed — Subject decision | 1 | 0 | 0
Not completed — Inclusion / Exclusion Criterion | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Primary Efficacy Analysis Set (24 week)
Groups:
- Apixaban (Primary SOC Information): Participants were treated with Apixaban 2.5 mg or 5 mg by mouth twice daily for 48 weeks and received Primary Standard of Care (SOC) information.
- Total: Total of all reporting groups
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program) | Total
Number analyzed (Participants) | 583 | 579 | 1162
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (8.94) | 73.1 (9.05) | 72.9 (9.00)
Age, Customized [Count of Participants; unit: Participants]
  <64 years | 86 | 77 | 163
  64-74 years | 221 | 220 | 441
  >=75 years | 276 | 282 | 558
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 234 | 466
  Male | 351 | 345 | 696

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With a Correct Execution of the Apixaban Dosing Regimen
Description: The mean percentage of days which participants maintained adherence to apixaban treatment was measured for each arm. Adherence to apixaban = number of units of adherence *100 / total number of eligible days for the time period from first dose date, up to 169 days. Unit of adherence: A 24-hour window where the treatment is taken as prescribed, ie, 1 tablet (5 mg or 2.5 mg, as appropriate) 2 times a day. If only one dose is missed in 24-hours, it is still considered as a unit of adherence. Adherence up to 24 weeks was calculated as the percentage of adherence units within that period. If a participant discontinued from the study before 24 weeks, the denominator time period was censored at the earlier of last dose date or discontinuation date for discontinuation due to reasons unrelated to participant adherence, such as withdrawn consent, or AE; otherwise, the period was censored at the minimum of 169 days and last dose date + 30 days.
Time Frame: Day 1 up to week 24
Population: Primary efficacy analysis set (Week 24), which consists of all randomized participants
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program)
Number analyzed (Participants) | 583 | 579
percentage of days | 91.64 (17.143) | 91.88 (16.140)
Statistical Analysis 1: Comparison: Apixaban (Primary SOC Information) vs Apixaban (Additional Educational Program); Test type: Superiority or Other; p = 0.8117, t-test, 2 sided — P-value (two-sided) corresponds to the two-sample t-tests for difference in percentage of adherence at Week 24; Difference in Percentage = -0.24, 95% CI 2-sided [-2.18 to 1.7]

2. Secondary Outcome: Percentage of Days With a Correct Execution of the Apixaban Dosing Regimen During the 12 to 24 Weeks Period Compared With During the First 12 Weeks
Description: The mean adherence to apixaban treatment during the first 24 weeks was measured between the standard of care (SOC) information and Additional Education Program (AEP) arms and expressed as a percentage. Adherence to Apixaban = number of units of adherence *100 / total number of eligible days for the time period.
Time Frame: Day 1 to Week 12, Week 12 to Week 24
Population: Primary efficacy analysis set (Week 24) with available data at both study days 85 and 169
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program)
Number analyzed (Participants) | 583 | 579
percentage
  Day 1 to Week 12: number analyzed (Participants) | 525 | 527
  Day 1 to Week 12 | 93.7 (14.18) | 93.0 (15.71)
  Week 12 to Week 24: number analyzed (Participants) | 525 | 527
  Week 12 to Week 24 | 90.3 (20.64) | 90.9 (18.36)
Statistical Analysis 1: Comparison: Apixaban (Primary SOC Information); Percent adherence at 12 Weeks v. Percent adherence at 24 Weeks; Test type: Superiority or Other; p < 0.0001, paired t-test — P-value is from a paired t-test comparing percent adherence at 12 and 24 Weeks. Only participants with available data at both Study Days 85 and 169 are included
Statistical Analysis 2: Comparison: Apixaban (Additional Educational Program); Percent adherence at 12 Weeks v. Percent adherence at 24 Weeks; Test type: Superiority or Other; p < 0.0001, paired t-test — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Days With a Correct Execution of the Apixaban Dosing Regimen During the 24 to 48 Weeks Period
Description: The mean percentage of days which participants maintained adherence to apixaban treatment was measured for each arm. Adherence to apixaban = number of units of adherence *100 / total number of eligible days for the time period from first dose date, up to 169 days. Unit of adherence: A 24-hour window where the treatment is taken as prescribed, ie, 1 tablet (5 mg or 2.5 mg, as appropriate) 2 times a day. If only one dose is missed in 24-hours, it is still considered as a unit of adherence. Adherence over 24 weeks was calculated as the percentage of adherence units within that period. If a participant discontinued from the study before 48 weeks, the denominator time period was censored at the earlier of last dose date or discontinuation date for discontinuation due to reasons unrelated to participant adherence, such as withdrawn consent, or AE; otherwise, the period was censored at the minimum of 169 days and last dose date + 30 days.
Time Frame: Week 24 to Week 48
Population: All treated participants in 24 to 48-week period. Participants that had not been using the EMD consistently throughout the study were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program) | Apixaban (Secondary SOC)
Number analyzed (Participants) | 510 | 253 | 254
percentage | 87.59 (22.921) | 88.41 (22.148) | 87.51 (21.125)
Statistical Analysis 1: Comparison: Apixaban (Primary SOC Information) vs Apixaban (Additional Educational Program) vs Apixaban (Secondary SOC); Test type: Non-Inferiority or Equivalence — F-test p-value is obtained from the one-way ANOVA model; p = 0.8707, ANOVA
Statistical Analysis 2: Comparison: Apixaban (Additional Educational Program) vs Apixaban (Secondary SOC); Test type: Superiority or Other; p = 0.6399, t-test, 2 sided — P-values are obtained from the Cochran t-test for pairwise comparison between groups (two-sided); Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-2.88 to 4.68]
Statistical Analysis 3: Comparison: Apixaban (Primary SOC Information) vs Apixaban (Secondary SOC); Test type: Superiority or Other; p = 0.9616, t-test, 2 sided — P-values are obtained from the Cochran t-test for pairwise comparison between groups (two-sided); Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-3.45 to 3.29]
Statistical Analysis 4: Comparison: Apixaban (Primary SOC Information) vs Apixaban (Additional Educational Program); Test type: Superiority or Other; p = 0.6341, t-test, 2 sided — P-values are obtained from the Cochran t-test for pairwise comparison between groups (two-sided); Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-2.60 to 4.24]

4. Secondary Outcome: Non-adherence Predictors of 20% or More (vs. at Least 80% Adherence) at 24 Weeks
Description: Logit analyses were conducted on the Primary Efficacy Set to identify non-adherence predictors of 20% or more (vs. at least 80% adherence) at 24 weeks. In the Primary SOC group, alcohol use, Mini-Mental State Evaluation (MMSE) score, UK standard occupational classification, and type of atrial fibrillation were retained in the model (p-value <= 0.2). In the Additional Educational Program group, alcohol use, type of atrial fibrillation, age and Vitamin K Antagonists (VKA) status were retained in the model (p-value <= 0.2). Odds ratios are presented for predictors of non-adherence.
Time Frame: Week 24
Population: Primary Efficacy Set participants with evaluable data at week 24
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program)
Number analyzed (Participants) | 557 | 560
Odds ratio
  <=2 Alcoholic Drink/Day Average vs None | 1.251 [0.691 to 2.265] | 0.994 [0.558 to 1.682]
  >=3 Alcoholic Drink/Day Average vs None | 4.268 [1.226 to 14.859] | 3.782 [0.884 to 16.178]
  Mini-mental state examination score | 0.808 [0.686 to 0.952] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Higher mgmt., adm. and professional jobs vs UKSOC1 | 0.827 [0.136 to 5.033] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Higher professional occupations vs UKSOC1 | 0.898 [0.197 to 4.091] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Intermediate occupations vs UKSOC1 | 1.230 [0.401 to 3.769] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Large employers and mgmt. and adm. jobs vs UKSOC1 | 2.823 [0.412 to 19.338] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Lower mgmt., adm. and professional jobs vs UKSOC1 | 0.948 [0.256 to 3.515] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Lower supervisory and tech. occupations vs UKSOC1 | 3.587 [1.008 to 12.766] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Never worked and long-term unemployed vs UKSOC1 | 1.289 [0.419 to 3.962] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Routine occupations vs UKSOC1 | 0.508 [0.181 to 1.425] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Semi-routine occupations vs UKSOC1 | 0.450 [0.083 to 2.453] | NA [NA to NA] — Not retained in model (p-value > 0.2)
  Paroxysmal vs Persistant Atrial Fibrillation | 1.626 [0.766 to 3.453] | 1.911 [0.940 to 3.885]
  Permanent vs Persistant Atrial Fibrillation | 2.560 [1.152 to 5.688] | 1.846 [0.819 to 4.158]
  VKA Naïve vs Non-Naïve | NA [NA to NA] — Not retained in model (p-value > 0.2) | 1.686 [0.932 to 3.049]
Statistical Analysis 1: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.1924, Wald Chi-square test — <=2 Drink/Day Average vs None
Statistical Analysis 2: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.0305, Wald Chi-square test — >=3 Drink/Day Average vs None
Statistical Analysis 3: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.0107, Wald Chi-square test — Mini-mental state examination score
Statistical Analysis 4: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.6982, Wald Chi-square test — Higher managerial, administrative and professional occupations vs UKSOC1
Statistical Analysis 5: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.7277, Wald Chi-square test — Higher professional occupations vs UKSOC1
Statistical Analysis 6: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.7581, Wald Chi-square test — Intermediate occupations vs UKSOC1
Statistical Analysis 7: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.2328, Wald Chi-square test — Large employers and higher managerial and adm. occupations vs UKSOC1
Statistical Analysis 8: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.7507, Wald Chi-square test — Lower managerial, administrative and professional occupations vs UKSOC1
Statistical Analysis 9: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.0091, Wald Chi-square test — Lower supervisory and technical occupations vs UKSOC1
Statistical Analysis 10: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.6730, Wald Chi-square test — Never worked and long-term unemployed vs UKSOC1
Statistical Analysis 11: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.0117, Wald Chi-square test — Routine occupations vs UKSOC1
Statistical Analysis 12: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.1910, Wald Chi-square test — Semi-routine occupations vs UKSOC1
Statistical Analysis 13: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.9559, Wald Chi-square test — Paroxysmal vs Persistent Atrial Fibrillation
Statistical Analysis 14: Comparison: Apixaban (Primary SOC Information); Test type: Superiority; p = 0.0264, Wald Chi-square test — Permanent vs Persistant Atrial Fibrillation
Statistical Analysis 15: Comparison: Apixaban (Additional Educational Program); Test type: Superiority; p = 0.1087, Wald Chi-square test — <=2 Drink/Day Average vs None
Statistical Analysis 16: Comparison: Apixaban (Additional Educational Program); Test type: Superiority; p = 0.0679, Wald Chi-square test — >=3 Drink/Day Average vs None
Statistical Analysis 17: Comparison: Apixaban (Additional Educational Program); Test type: Superiority; p = 0.2128, Wald Chi-square test — Paroxysmal vs Persistant Atrial Fibrillation
Statistical Analysis 18: Comparison: Apixaban (Additional Educational Program); Test type: Superiority; p = 0.3739, Wald Chi-square test — Permanent vs Persistant Atrial Fibrillation
Statistical Analysis 19: Comparison: Apixaban (Additional Educational Program); Test type: Superiority; p = 0.843, Wald Chi-square test — VKA status: Naive vs. Non-Naive

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Drug Related Adverse Events (AE), AE Leading to Discontinuation, and Death
Description: AEs with onset date from day 1 through week 24 are included in this summary. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Day 1 up to week 24
Population: All randomized participants. Participants in the safety analysis set were categorized according to the counseling actually received
Measure: Number; unit: Participants
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program)
Number analyzed (Participants) | 604 | 558
Participants
  SAE | 75 | 82
  Drug related AE | 54 | 41
  AE leading to discontinuation | 33 | 22
  Death | 6 | 5

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Drug Related Adverse Events (AE), AE Leading to Discontinuation, and Death
Description: Adverse events with onset date after 24 weeks are included in this summary. AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Week 24 up to Week 48
Population: All randomized participants remaining in the study after week 24. All randomized participants. Participants in the safety analysis set were categorized according to the counseling actually received
Measure: Number; unit: Participants
Arm/Group | Apixaban (Primary SOC Information) | Apixaban (Additional Educational Program) | Apixaban (Secondary SOC)
Number analyzed (Participants) | 604 | 308 | 223
Participants
  SAE | 71 | 43 | 30
  Drug related AE | 15 | 12 | 10
  AE leading to discontinuation | 14 | 3 | 8
  Death | 3 | 3 | 6

ADVERSE EVENTS:
Time Frame: From date of first dose to date of last dose plus 30 days
Description: All randomized participants were analyzed. Participants in the safety analysis set were categorized according to the counseling actually received.
Groups:
- Primary SOC (Period 1): Apixaban 2.5 mg or 5 mg by mouth twice daily for 24 weeks and Primary SOC information.
- Continued Additional Educational Program (CAEP) (Period 2): Subjects enrolled in AEP program during the first 24 weeks continued receiving AEP program up to 48 weeks.
- Secondary SOC (Period 2): Subjects who received AEP for 24 weeks then revert to SOC after the second randomization.
- Additional Educational Program (Period 1): Apixaban 2.5 mg or 5 mg by mouth twice daily for 24 weeks and Additional Educational Program.
- Primary SOC (Period 2): Subjects who received Apixaban 2.5 mg or 5 mg by mouth twice daily for initial 24 weeks and Primary SOC information continued for a period 48 Weeks.
Arm/Group | Primary SOC (Period 1) | Continued Additional Educational Program (CAEP) (Period 2) | Secondary SOC (Period 2) | Additional Educational Program (Period 1) | Primary SOC (Period 2)
Serious Adverse Events (participants affected / at risk) | 69/604 | 40/308 | 29/223 | 79/558 | 62/604
Other Adverse Events (participants affected / at risk) | 40/604 | 5/308 | 5/223 | 46/558 | 21/604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary SOC (Period 1) (N=604) | Continued Additional Educational Program (CAEP) (Period 2) (N=308) | Secondary SOC (Period 2) (N=223) | Additional Educational Program (Period 1) (N=558) | Primary SOC (Period 2) (N=604)
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Arthroscopic surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Breast conserving surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 8 | 1 | 0 | 3 | 3
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 1
Cardioversion (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Corneal transplant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Coronary artery bypass (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
Heart valve replacement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0 | 0 | 2 | 0
Intervertebral disc operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Lung lobectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 0 | 0 | 2 | 0
Spinal operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Scar excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Vascular graft (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Elderly (Social circumstances) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 1 | 3
Drug intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Implant site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Multi-Organ failure (General disorders) | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Aspiration breast (Investigations) | 0 | 1 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 0 | 0 | 1 | 0 | 1
Blood test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy lung (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Catheterisation cardiac (Investigations) | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2 | 1 | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 2 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 0 | 1 | 10 | 3
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 9 | 3 | 1 | 13 | 4
Cardiac flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Post stroke seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 3 | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Diabetic gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 1 | 2 | 3 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Streptococcal endocarditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary SOC (Period 1) (N=604) | Continued Additional Educational Program (CAEP) (Period 2) (N=308) | Secondary SOC (Period 2) (N=223) | Additional Educational Program (Period 1) (N=558) | Primary SOC (Period 2) (N=604)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 5 | 5 | 46 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.